CLINICAL TRIAL: NCT03172377
Title: Lengthening Adalimumab Dosing Interval in Quiescent Crohn's Disease Patients
Acronym: LADI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: Erasmus Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL58948.091.16; 848015002 (Other Grant/Funding Number: ZonMW); 2016-003321-42 (EudraCT Number)
Record Dates: First submitted 2017-05-29; First posted 2017-06-01 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2021-11

CONDITIONS: Crohn Disease in Remission; Crohn Disease
Keywords: adalimumab; anti-tumor necrosis factor; anti-TNF; Humira; interval lengthening; dosing interval; inflammatory bowel disease; antidrug antibodies; trough levels; pharmacokinetics; immunogenicity; cost-effectiveness; dose reduction
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases

STUDY DESIGN:
Intervention Model Description: Multicenter, randomized controlled, open label non-inferiority trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Lengthening adalimumab dosing interval: The adalimumab injection interval during maintenance therapy (40 mg sc / 2 weeks) will be extended through a stepwise disease activity guided manner to 3 weeks and subsequently - after 24 weeks - to 4 weeks. If a step-down leads to recurrence of disease activity patients will return to the preceding effective dosing interval.
  Interventions: Other: Lengthening adalimumab dosing interval
- Control group (No Intervention): Standard care: patients will continue adalimumab maintenance treatment of 40mg per 2 weeks. Treatment decisions are made at the discretion of the treating physician.

INTERVENTIONS:
Other: Lengthening adalimumab dosing interval — Lengthening adalimumab dosing interval from 2 weeks to 3 weeks and -later- to 4 weeks.
  Other Names: Lengthening Humira dosing interval; Longer adalimumab interval; Longer Humira interval; Adalimumab dose reduction; Humira dose reduction
  Arms: Intervention group

SUMMARY:
Crohn's disease is a chronic inflammatory bowel disease. This disease can be treated with, among other things, biologicals such as adalimumab. Patients use adalimumab for a long time to maintain remission and to prevent relapse of the bowel inflammation. The disadvantages of this therapy are the high price and side effects (such as the higher risk of infection).

Currently, adalimumab is given every 2 weeks, by injection under the skin. The optimal time between two injections has never been investigated before. Prior research in patients with rheumatoid arthritis shows that disease remission can be maintained with longer injection-intervals. Our hypothesis is that this is the same for Crohn's disease patients. Our aim is to show non-inferiority of extending the adalimumab dosing interval, under strict disease monitoring in Crohn's disease patients in sustained (>9 months) clinical remission, compared to standard care.

During the trial,174 patients with stable Crohn's disease will be divided into 2 groups. One group continues adalimumab injections with the same 2-week interval. And the other group will incrementally extend the interval to 4 weeks, under strict disease monitoring. If a step-down leads to recurrence of disease activity patients will return to the preceding effective dosing interval. Thus, we will investigate whether, and for whom, it is safe to extend the adalimumab injection interval.

DETAILED DESCRIPTION:
Rationale

Adalimumab is both an effective induction and maintenance therapy for Crohn's disease (CD). Due to the risk of side effects (infections, injection reaction) and high costs, an extension of the injection interval is an attractive option. However, this strategy has not been evaluated yet in a randomized controlled trial in CD patients.

Objective

To assess non-inferiority and cost-effectiveness of disease activity guided adalimumab interval lengthening in CD patients in sustained (>9 months) clinical remission, compared to standard dosing of every other week.

Study design

Multicenter, randomized controlled, open label non-inferiority trial, with two treatment arms.

Study population

Crohn's disease patients, in sustained clinical remission on adalimumab maintenance therapy.

Intervention

Intervention arm: The adalimumab injection interval during maintenance therapy (40 mg per 2 weeks) will be extended through a stepwise disease activity guided manner to 3 weeks and subsequently - after 24 weeks - to 4 weeks. If a step-down leads to recurrence of disease activity patients will return to the preceding effective dosing interval.

Control arm: patients will continue adalimumab maintenance treatment of 40mg per 2 weeks. Treatment decisions are made at the discretion of the treating physician.

Main study parameters/endpoints

Primary outcome: Cumulative incidence of persistent disease flares in 48 weeks of follow-up. A persistent flare is defined as two of three of the following criteria persisting for > 8 weeks, despite dose escalation of adalimumab; FC >250 µg/g, CRP≥10 mg/L, HBI ≥5. Non-inferiority is reached if the difference in cumulative incidence of persistent flares not exceeds the non-inferiority margin of 15%.

Secondary outcomes include cumulative incidence of transient flares, adverse events, predictors for successful dose reduction and cost-effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of colonic and/or distal ileal CD
* Sustained steroid-free clinical remission for >9 months whilst being treated with adalimumab at a stable dose
* Adalimumab dosed at 40 mg sc every 2 weeks
* Full clinical response and disease control, all three criteria below need to be fulfilled prior to enrollment:

  * Absence of active inflammatory intestinal or extra-intestinal symptoms, as judged by both patient and physician
  * Fecal calprotectin (FC) < 150 μg/g and C reactive protein (CRP) <10 mg/L
  * Harvey Bradshaw Index (HBI) <5

Exclusion Criteria:

* Absence of written informed consent
* Concomitant corticosteroid usage
* Need for CD-related surgery
* Actively draining peri-anal fistula
* Pregnancy or lactation
* Other significant medical conditions that might interfere with this study (such as current/recent malignancy, immunodeficiency syndromes and psychiatric illness)
* Impossibility to measure outcomes, e.g. planned relocation, language issues, short life expectancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2017-05-03 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of persistent disease flares. | From the date of randomization up to week 48.
  A persistent flare is defined as two of three of the following criteria persisting for > 8 weeks, despite dose escalation of adalimumab; FC >250 µg/g, CRP≥10 mg/L, HBI ≥5. Non-inferiority is reached if the difference in cumulative incidence of persistent flares not exceeds the non-inferiority margin of 15%.

SECONDARY OUTCOMES:
Cumulative incidence of transient disease flares. | From the date of randomization up to week 48.
  A transient flare is defined as two of three of the following criteria persisting for ≤ 8 weeks; FC >250 µg/g, CRP≥10 mg/L, HBI ≥5.
(Serious) adverse event rate | From the date of randomization up to week 48.
  (Serious) adverse events that are (possibly) related to adalimumab and the (Serious) adverse events that are (possibly) related to adalimumab interval lengthening in the intervention and control group, expressed as events/ 100 patient-years of follow-up.
Whether adalimumab drug level is associated with successful interval lengthening | From the date of randomization up to week 48.
  Adalimumab drug levels at baseline measured by ELISA.
Whether biochemic FC or CRP are associated with successful interval lengthening | From the date of randomization up to week 48.
  Fecal calprotectin (mg/kg) or C-reactive protein (mg/L).
Whether co-medication use is associated with successful interval lengthening | From the date of randomization up to week 48.
  Co-medication includes azathioprine, Co-medication includes azathioprine, 6-mercaptopurine, 6-thioguanine, methotrexate.
The decremental cost effectiveness ratio of this interval lengthening strategy | From the date of randomization up to week 48.
  Dividing the difference in costs (based on medical consumption (by medical consumption questionnaire(MCQ)) and work productivity (by productivity cost questionnaire(PCQ))) by the difference in quality-adjusted life years (based on EuroQol-5D questionnaire).

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Hoentjen, MD, PhD, Principal Investigator — Radboud University Medical Center; Prof. dr. van der Woude, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (22):
- Netherlands (22):
  - Radboudumc University Nijmegen Medical Centre, Nijmegen, Gelderland
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch, North Brabant
  - Amphia Ziekenhuis, Breda, North Brabant
  - Bernhoven, Uden, North Brabant
  - VU Medisch Centrum, Amsterdam, North Holland
  - Albert Schweitzer Ziekenhuis, Dordrecht, South Holland
  - Franciscus Gasthuis & Vlietland, Rotterdam, South Holland
  - Erasmus Medical Center, Rotterdam, South Holland
  - Ikazia Ziekenhuis, Rotterdam, South Holland
  - Flevoziekenhuis, Almere Stad
  - AmsterdamUMC - location AMC, Amsterdam
  - Onze Lieve Vrouwe Gasthuis (OLVG), Amsterdam
  - Reinier de Graaf, Delft
  - Maxima Medisch Centrum, Eindhoven
  - Medisch Spectrum Twente, Enschede
  - Zuyderland ziekenhuis, Geleen
  - Spaarne Gasthuis, Haarlem
  - Leids Universitair Medisch Centrum, Leiden
  - Maastricht UMC+, Maastricht
  - Canisius Wilhelmina Ziekenhuis, Nijmegen
  - Elisabeth-TweeSteden Ziekenhuis, Tilburg
  - UMC Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] van Linschoten RCA, Jansen FM, Pauwels RWM, Smits LJT, Atsma F, Kievit W, de Jong DJ, de Vries AC, Boekema PJ, West RL, Bodelier AGL, Gisbertz IAM, Wolfhagen FHJ, Romkens TEH, Lutgens MWMD, van Bodegraven AA, Oldenburg B, Pierik MJ, Russel MGVM, de Boer NK, Mallant-Hent RC, Ter Borg PCJ, van der Meulen-de Jong AE, Jansen JM, Jansen SV, Tan ACITL, van der Woude CJ, Hoentjen F; LADI study group, the Dutch Initiative on Crohn, Colitis (ICC). A Prediction Model for Successful Increase of Adalimumab Dose Intervals in Patients with Crohn's Disease: Secondary Analysis of the Pragmatic Open-Label Randomised Controlled Non-inferiority LADI Trial. Dig Dis Sci. 2024 Jun;69(6):2165-2174. doi: 10.1007/s10620-024-08410-z. Epub 2024 Apr 9. PMID 38594435
- [Derived] Jansen FM, van Linschoten RCA, Kievit W, Smits LJT, Pauwels RWM, de Jong DJ, de Vries AC, Boekema PJ, West RL, Bodelier AGL, Gisbertz IAM, Wolfhagen FHJ, Romkens TEH, Lutgens MWMD, van Bodegraven AA, Oldenburg B, Pierik MJ, Russel MGVM, de Boer NK, Mallant-Hent RC, Ter Borg PCJ, van der Meulen-de Jong AE, Jansen JM, Jansen SV, Tan ACITL, Hoentjen F, van der Woude CJ; LADI study group. Cost-Effectiveness Analysis of Increased Adalimumab Dose Intervals in Crohn's Disease Patients in Stable Remission: The Randomized Controlled LADI Trial. J Crohns Colitis. 2023 Nov 24;17(11):1771-1780. doi: 10.1093/ecco-jcc/jjad101. PMID 37310877
- [Derived] van Linschoten RCA, Jansen FM, Pauwels RWM, Smits LJT, Atsma F, Kievit W, de Jong DJ, de Vries AC, Boekema PJ, West RL, Bodelier AGL, Gisbertz IAM, Wolfhagen FHJ, Romkens TEH, Lutgens MWMD, van Bodegraven AA, Oldenburg B, Pierik MJ, Russel MGVM, de Boer NK, Mallant-Hent RC, Ter Borg PCJ, van der Meulen-de Jong AE, Jansen JM, Jansen SV, Tan ACITL, van der Woude CJ, Hoentjen F; LADI study group and the Dutch Initiative on Crohn and Colitis. Increased versus conventional adalimumab dose interval for patients with Crohn's disease in stable remission (LADI): a pragmatic, open-label, non-inferiority, randomised controlled trial. Lancet Gastroenterol Hepatol. 2023 Apr;8(4):343-355. doi: 10.1016/S2468-1253(22)00434-4. Epub 2023 Jan 31. PMID 36736339
- [Derived] Smits LJT, Pauwels RWM, Kievit W, de Jong DJ, de Vries AC, Hoentjen F, van der Woude CJ; LADI study group. Lengthening adalimumab dosing interval in quiescent Crohn's disease patients: protocol for the pragmatic randomised non-inferiority LADI study. BMJ Open. 2020 May 26;10(5):e035326. doi: 10.1136/bmjopen-2019-035326. PMID 32461297
- See also: Dutch organisation for healthcare research and innovation (ZonMW) — https://www.zonmw.nl/nl/over-zonmw/innovatie-in-de-zorg/programmas/project-detail/goed-gebruik-geneesmiddelen/lengthening-adalimumab-dosing-interval-in-quiescent-crohns-disease-patients-the-ladi-study/